CLINICAL TRIAL: NCT02233621
Title: Evaluation Des Performances de la Tomographie Par Emission de Positons Avec la 16α-[18F]Fluoro-17β-estradiol ([18F]-FES) Pour le Diagnostic de l'Endometriose
Brief Title: Assessment of Performance of [18F]-FES for Endometriosis Diagnosis
Acronym: ENDOTEP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: not enough enrollement
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 49RC10_32_01-PHRC2010-02; 2011-003734-14 (EudraCT Number)
Record Dates: First submitted 2014-08-29; First posted 2014-09-08 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2014-09

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — 16-fluoroestradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PET with [18F]-FES (Experimental): PET with [18F]-FES compared to histological analysis performed at least on one biopsy done during coelioscopy.
  Interventions: Other: [18F]FES (16α-[18F]Fluoro-17β-estradiol)

INTERVENTIONS:
Other: [18F]FES (16α-[18F]Fluoro-17β-estradiol) — PET with [18F]FES before coelioscopy
  Other Names: analog of estrogene

SUMMARY:
Endometriosis is a benign chronic disease responsible for infertility and pelvic pain. One of the main problem of endometriosis is the significant delay of diagnosis.This delay has significant consequences for patients. Currently the definitive diagnosis of endometriosis and the evaluation of its lesional extension require performing laparoscopy and a histological analysis of biopsy and pathologic areas. Lesions of endometriosis whose development and growth are estrogen-dependent, express estrogen receptor (ER). [18F]FES (16α-[18F]Fluoro-17β-estradiol) is an analog of estrogen, used in positron emission tomography (PET), and a specific tracer of ER. We propose to evaluate the performance of this functional imaging as a diagnostic tool for endometriosis.

The aim of this multicenter, prospective, open study is to assess sensitivity of PET with [18F] -FES for diagnosing endometriosis compared to the gold standard (histological confirmation on biopsy or excision of lesions performed during laparoscopy) in women care for suspected endometriosis and for whom laparoscopy is already scheduled.

ELIGIBILITY:
Inclusion Criteria:

* First planned coelioscopy (therapeutic indication) for suspected endometriosis
* Patient aged from 18 to 50 years
* Absence of treatment with GnRH (gonadotropin-releasing hormone) analogue for at least 3 months
* Patient affiliated to a social security system
* No hormonal treatment for at least 3 months

Exclusion Criteria:

* History of abdominal pelvic surgery for endometriosis
* Current treatment with GnRH (gonadotropin-releasing hormone) or stopped for less than 3 months
* hormonal Drug ongoing
* Patient pregnant, may be or during lactation
* Patient under guardianship or trusteeship
* Patient unable to understand the purpose of the study
* Patient already included in another clinical trial with an experimental molecule.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2012-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04-06

PRIMARY OUTCOMES:
sensitivity of PET with [18F] -FES for diagnosing endometriosis defined by the ability of this diagnostic exam to give a positive result when endometriosis is present | Within 3 months after inclusion when laparoscopy is already scheduled.
  PET with [18F]-FES considered positive if it allows to identify at least one hyperfixation area in a physiologically area not fixing tracer or not corresponding to a physiological removal area tracer.
  PET results will be correlated with The results of PET with [18F] -FES will be correlated with histology results of at least one of the biopsies performed at laparoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Descamps, PU-PH, Study Chair — University Hospital of Angers; Olivier Couturier, PU-PH, Principal Investigator — University Hospital of Angers; Céline Lefebvre-Lacoeuille, PH, Principal Investigator — University Hospital of Angers
Locations (1):
- Nuclear medicin unit, University Hospital of Angers, Angers, France